CLINICAL TRIAL: NCT01420042
Title: A Phase I, Double-Blind, Randomized, Dose Escalation Study to Assess the Safety, Tolerability, and Pharmacokinetics of NNZ-2566 in Healthy Subjects, Following Oral Administration
Brief Title: Safety Study of NNZ-2566 in Healthy Subjects, Following Oral Administration
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Neuren Pharmaceuticals Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Neu-2566-HV-005
Record Dates: First submitted 2011-08-17; First posted 2011-08-19 (Estimated); Last update posted 2012-11-22 (Estimated); Status verified 2012-11

CONDITIONS: Brain Injuries, Traumatic
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — trofinetide; Water; Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (lemon flavoured cordial) (Placebo Comparator): NNZ-2566 reconstituted in Lemon flavoured cordial and Water for Injection. 6/8 subjects in each cohort (3 cohorts in total) to receive NNZ-2566 experimental treatment.
  Interventions: Drug: Placebo
- NNZ-2566 (Experimental)
  Interventions: Drug: NNZ-2566

INTERVENTIONS:
Drug: NNZ-2566 — Glycyl-L-2-Methylprolyl-L-Glutamic Acid (NNZ-2566) supplied as a lyophilized powder (2g in 50mL vials) for reconstitution with lemon flavoured cordial and Water for Injection.
  Other Names: NNZ-2566 Lot NNZP25
  Arms: NNZ-2566
Drug: Placebo — Lemon flavoured cordial and Water for Injection
  Other Names: Bickford's Bitter Lemon Cordial, 1:1 in Water for Injection
  Arms: Placebo (lemon flavoured cordial)

SUMMARY:
The purpose of this study is to obtain evidence of safety and determine the pharmacokinetics (PK) of NNZ-2566 in healthy volunteers, when administered orally.

DETAILED DESCRIPTION:
Double-blind, placebo-controlled, randomized (with a 6:2 randomization for active versus placebo) safety, dose-escalation, and pharmacokinetic study of NNZ-2566.

Three cohorts will be sequentially dosed, starting with two cohorts receiving a single dose (6mg/kg followed by 30mg/kg). The third cohort will receive two 100mg/kg doses over the course of one day and following a formal safety review the same subjects will then receive two 100mg/kg doses each day for five days.

ELIGIBILITY:
Inclusion Criteria:

* Males: 60.0-100.0 kg, Females: 50.0-100.0 kg (inclusive).
* Males: Body mass index (BMI) of 20-30.0, Females: BMI of 18.5-30.0 kg/m2 (inclusive).
* Healthy, determined by a medical history with particular attention to:

  * drug history identifying any known drug allergies and the presence of drug abuse;
  * any chronic use of medication
  * thorough review of body systems: no clinically significant abnormal findings on physical examination and electrocardiogram (ECG),
* Adequate venous access in arms to allow collection of blood samples.
* Fluent in the English language.
* Have voluntarily given written informed consent.

Exclusion Criteria:

* Pregnant and lactating females.
* History of allergy/hypersensitivity to any of the ingredients of the formulations
* History of clinically significant gastrointestinal, hepatic, renal, cardiovascular, dermatological, immunological, respiratory, endocrine, oncological, neurological, metabolic, gynecological, ENT or musculoskeletal disorders, psychiatric disease or hematological disorders.
* Any history of asthma during the last 10 years.
* Creatinine clearance <65 mL/min.
* Any predisposing condition that might interfere with the absorption, distribution, metabolism, and/or excretion of the investigational product.
* History of abnormal bleeding tendencies or thrombophlebitis unrelated to venepuncture.
* History of hepatitis B, a positive test for hepatitis B surface antigen, a history of hepatitis C, a positive test for hepatitis C antibody, a history of HIV infection or demonstration of HIV antibodies.
* Any evidence of organ dysfunction, or any clinically significant clinical laboratory value which, in the opinion of the Investigator would jeopardize the safety of the subject or impact on the validity of the study results, including a liver function test (LFT) >1.5 x upper limit of normal (ULN).
* Those who may have difficulty abstaining from alcohol during the 48 hr prior to dose administration and until completion of the Study Exit visit.
* History of, or current evidence of, abuse of alcohol or any drug substance, licit or illicit, or positive urine drug screen for drugs of abuse.
* Difficulty in abstaining from any prescription medications for 14 days prior to dose administration and for the duration of the study.
* Difficulty in abstaining from over-the-counter (OTC) medications or herbal supplements for 14 days prior to dose administration and for the duration of the study, (with the exception of occasional analgesia, vitamin and other nutrient supplement use, at the discretion of the Investigator).
* Difficulty in abstaining from food and/or beverages that contain caffeine or other xanthines, (e.g. coffee, tea, cola and chocolate) during the 48 hrs prior to dose administration and for the duration of the study.
* History of any psychiatric illness which may impair the ability to provide written informed consent.
* Poor compliers or those unlikely to attend.
* Receipt of any drug as part of a research study within 30 days of initial dose administration in this study.
* Standard blood donation (usually 550 mL) within the 12-week period before dose administration.
* Unusual dietary habits and excessive or unusual vitamin intakes.
* Vaccination or immunizations within 30 days of initial dose administration.
* Whilst there were no QT/QTc effects seen in the human volunteers at a dose of 20 mg/kg administered intravenously as a 10 min infusion, until the effects of the drug on QT/QTc interval have been formally characterized, the study will use the exclusion criteria defined in International Conference on Harmonisation (ICH) Guideline E14 to exclude subjects with a risk of QT/QTc prolongation, namely:

  * A marked baseline prolongation of corrected QT interval >450 ms in two ECGs, or
  * A history of risk factors for Torsade de Pointes (e.g., heart failure, hypokalemia, family history of Long QT Syndrome).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2012-02; Primary Completion 2012-08 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events (AE) and serious adverse events (SAE) | Through to Day 7 post end of study drug administration or until resolved

CONTACTS AND LOCATIONS:
Overall Officials: Maggie Scott, Principal Investigator — Neuren Pharmaceuticals Ltd
Locations (1):
- Nucleus Network, Melbourne, Victoria, Australia